CLINICAL TRIAL: NCT04757181
Title: Influence of Diet on Microbiome and Inflammation
Brief Title: The Inflammatory Bowel Disease - Anti-Inflammatory Diet (IBD-AID)
Acronym: IBD-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Ana Maldonado-Contreras, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00008033
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The study design is a single-arm, prospective, pre-post intervention trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBD patients (Experimental): IBD patients will be used as their own control. Participants will start the study in a baseline phase (4 weeks) and intervention phase (8 weeks)
  Interventions: Other: The IBD-AID

INTERVENTIONS:
Other: The IBD-AID — Subjects will meet with study personnel for to fill out baseline questionnaires (approximately a 1-hour visit). Subjects will be instructed to make dietary changes based one the IBD-AID guidelines. Dietary instruction will be delivered via individual and group sessions led by trained study personnel. Participants will be expected to learn the skills of dietary change to the IBD-AID and will begin their 8 weeks compliance period followed by endpoint measures. Participants are encouraged to attend 3 cooking classes (1.5 hours duration) in our teaching kitchen.

SUMMARY:
The goal of this study is to prospectively test the hypothesis that specific dietary modification can improve patient symptoms by promoting beneficial changes in the composition of the microbiome that, in turn, alter the immune response in such a way as to and ameliorate inflammatory conditions such as Inflammatory Bowel Disease (IBD). The potential long term benefit of this research is a validated set of efficacious dietary guidelines for persons with IBD. The potential immediate benefit to patients is symptomatic relief and healing.

DETAILED DESCRIPTION:
The gut microbiome is the community of microbes that inhabit the gastrointestinal tract. Sequencing and analysis of the DNA and/or RNA of the gut microbiome (metagenomics) allow the identification of the species present and assess the metabolic activities they carry out. Stools are largely microbial and the metagenomics of stool can provide insights into the functioning of the gut microbiome.

Nutrient processing by the gut microbiome is fundamental to energy extraction and immune response. Until recently, investigation of nutritional approaches to treating Inflammatory bowel diseases (IBD) has been largely limited to the use of enteral and total parenteral nutrition with the aim of providing bowel rest.

The IBD Anti-inflammatory diet (IBD-AID) was developed to establish a dietary therapy to address nutritional adequacy and malabsorption issues, promote symptom relief, and assist with remission. The IBD-AID has been designed to favor colonic bacteria that degrade dietary fibers and produce short-chain fatty acids (SCFAs). SCFAs regulate the production of cytokines (TNF-α, IL-2, IL-6, and IL-10), eicosanoids, and chemokines (e.g., MCP-1 and CINC-2) by acting on macrophages and endothelial cells. High levels of SCFAs then promote a hyporesponsive immunological environment to commensal bacteria through the down-regulation of those pro-inflammatory effectors, aiding homeostasis maintenance.

This diet utilizes foods that are available in most grocery stores and is intended to be a complete diet that provide balanced nutrition. As many of the available medical treatments for inflammatory bowel disease have risks, this diet may be a safer alternative to medical treatment in this population. The nutrition recommendations are safe. Diet modification poses minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* - 15 years of age or older
* Willingness and capacity to significantly change diet
* Willing and able to comply with scheduled visits, blood, and stool collection, and other study procedures and to complete the study
* Clinical provider (GI clinician) permission for IBD patients to participate in the intervention is required for participation in the study.
* Evidence of personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* For children age 15 and above, the assent of the child and consent of a parent or legal guardian will be required.
* One of the following:

  * diagnosis of IBD, specifically Crohn's Disease and Ulcerative Colitis
  * healthy control

Exclusion Criteria:

* the presence of infection (such as C.diff) precipitating the colitis
* antibiotics taken within 3 months of study entry
* medically unstable to give consent
* on heparin or Coumadin
* Prisoners
* Subjects who do not speak or understand English, to ensure that there is consistency in teaching and educational materials.
* Subjects who self-report current pregnancy
* Patients who do not receive clinical care at UMass Memorial Health Care

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Microbiome change after the IBD-AID | 8 weeks
  Analysis of the microbial composition of the gut and changes that correlate with diet compliance

SECONDARY OUTCOMES:
Improvement of symptoms | 8 weeks
  Assessment of disease severity and overall quality of life before and after the IBD-AID
Improvement of inflammatory markers | 8 weeks
  Assessment of inflammatory markers in blood before and after the IBD-AID

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No